CLINICAL TRIAL: NCT03043651
Title: An Open-label Extension Study of Oral Treprostinil in Subjects With Pulmonary Hypertension (PH) Associated With Heart Failure With Preserved Ejection Fraction (HFpEF) - A Long-term Follow-up to Study TDE-HF-301
Brief Title: Open-label Extension of Oral Treprostinil in Subjects With PH Associated With HFpEF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-HF-302
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Hypertension Associated With HFpEF
Keywords: Pulmonary Hypertension; HFpEF; 6-Minute Walk Test; Oral Treprostinil
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral treprostinil (Experimental): Sustained-release tablets for TID administration
  Interventions: Drug: Oral treprostinil

INTERVENTIONS:
Drug: Oral treprostinil — Sustained-release oral tablets for TID administration
  Other Names: Treprostinil diethanolamine, Treprostinil diolamine

SUMMARY:
This was an open-label study to evaluate the safety of continued therapy with oral treprostinil in subjects who completed Study TDE-HF-301. This study provided long-term, open-label data regarding the effect of continued long-term oral treprostinil therapy for the treatment of pulmonary hypertension (PH) associated with heart failure with preserved ejection fraction (HFpEF). Subject visits occurred at Baseline, Weeks 6, 12, 18, 24, and every 12 weeks thereafter until either oral treprostinil was commercially available to treat PH associated with HFpEF or the study was discontinued by the Sponsor.

The Sponsor terminated Studies TDE-HF-301 and TDE-HF-302 on 14 October 2019 due to slow enrollment. Safety data from the final subject in Study TDE-HF-302 were recorded on 02 March 2020. Due to the lower than expected number of subjects enrolled, the planned secondary efficacy-related endpoints were not analyzed.

DETAILED DESCRIPTION:
Study TDE-HF-302 was a multicenter, open-label study in subjects participating and completing all required visits for Study TDE-HF-301. This study assessed the long-term safety of oral treprostinil in subjects with PH associated with HFpEF.

Subjects received oral treprostinil as 0.125-, 0.25-, 1-, and 2.5-mg sustained-release tablets. For subjects who were randomly allocated to receive oral treprostinil in Study TDE-HF-301, the initial dose of oral treprostinil was the same as the final dose in Study TDE-HF-301. Subjects randomly allocated to receive placebo in Study TDE-HF-301 were administered the initial dose of oral treprostinil at 0.125 mg 3 times daily (TID). Dose increases could occur in 0.125-mg increments every 72 hours at the discretion of the Investigator up to 6 mg TID, the maximum allowable dose determined by the Data Monitoring Committee during Study TDE-HF-301. Doses of study drug were to be increased in the absence of dose-limiting drug-related adverse events (AEs) to ensure that each subject received the optimal dose throughout the study. Subjects returned for visits at Weeks 6, 12, 18, and 24, and every 12 weeks thereafter. Subjects who terminated the study early were asked to return to the study center for a final evaluation.

Safety assessments consisted of AEs, clinical laboratory parameters, and clinical assessment of heart failure signs and symptoms.

Due to the lower than expected number of subjects enrolled, the planned secondary efficacy-related endpoints were not analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. The subject participated in Study TDE-HF-301, remained on study drug, was compliant with study procedures and assessments during Study TDE-HF-301, and completed through Week 24 of that study.

Exclusion Criteria:

1. The subject was pregnant or lactating.
2. The subject was prematurely discontinued from Study TDE-HF-301 for any reason.
3. The subject developed a concurrent illness or condition during Study TDE-HF-301, which, in the opinion of the Investigator, represented a risk to the subject's overall health if they enrolled in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Gomberg-Maitland, MD, Principal Investigator — George Washington University
Locations (82):
- United States (82):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - VA Healthcare System of Greater Los Angeles, Los Angeles, California
  - University of California Los Angeles Pulmonary Division, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - South Denver Cardiology, Littleton, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medical Faculty Associates, George Washington University, Washington D.C., District of Columbia
  - Bay Area Cardiology Associates, Brandon, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - St. Vincent's Lung, Sleep, and Critical Care Specialists, Jacksonville, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - University of South Florida ; Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic of Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Piedmont Physicians Georgia Lung, Austell, Georgia
  - WellStar Medical Group, Marietta, Georgia
  - University of Illinois at Chicago Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - OSF HealthCare, Peoria, Illinois
  - Indiana University Health Methodist Research Institute, INC, Indianapolis, Indiana
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville Physicians Outpatient Center, Louisville, Kentucky
  - Chest Medicine Associates, South Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Barnabas Health Lung Center, Newark, New Jersey
  - Albany Medical College, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Pulmonary Health Physicians, PC, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - The Lindner Research Center The Christ Hospital Health Network, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Toldedo Medical Center, Toledo, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AnMed Health Pulmonary and Sleep Medicine, Anderson, South Carolina
  - VitaLink Research - Anderson, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Summit Medical Group, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Providence Medical Research Center, Spokane, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Treprostinil
Started | 48
Completed | 0
Not Completed | 48
Not completed — Death | 1
Not completed — Progressive Disease | 2
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Study Terminated by Sponsor | 39

BASELINE CHARACTERISTICS:
Population: All Subjects
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 76.0 [46 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety of Oral Treprostinil in Subjects With PH Associated With HFpEF for Subjects Who Completed Study TDE-HF-301
Description: The primary objective of this study was to evaluate the long-term safety of oral treprostinil in subjects with PH associated with HFpEF for subjects who completed Study TDE-HF-301. The number of subjects with adverse events during the study is reported as the primary outcome measure, which was the only outcome measurement reported for this Sponsor-terminated study.
Time Frame: Baseline through study completion, up to approximately 25 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 48
Participants | 47

ADVERSE EVENTS:
Time Frame: The study duration was 25 months overall. The study was discontinued by the Sponsor on 14 October 2019 due to slow enrollment in the parent study, TDE-HF-301.
Arm/Group | Oral Treprostinil
All-Cause Mortality (participants affected / at risk) | 1/48
Serious Adverse Events (participants affected / at risk) | 19/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil (N=48)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Cardiac failure (Cardiac disorders) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia (Infections and infestations) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Death (General disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil (N=48)
Headache (Nervous system disorders) | 31 (35)
Diarrhoea (Gastrointestinal disorders) | 26 (28)
Nausea (Gastrointestinal disorders) | 17 (20)
Fatigue (General disorders) | 15 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (20)
Dizziness (Nervous system disorders) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Oedema peripheral (General disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 5 (7)
Blood creatinine increased (Investigations) | 5 (5)
Chest pain (General disorders) | 5 (6)
Flushing (Vascular disorders) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5)
Pneumonia (Infections and infestations) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Hypotension (Vascular disorders) | 4 (5)
Oedema (General disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Cardiac failure (Cardiac disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 3 (3)
Palpitations (Cardiac disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Presyncope (Nervous system disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the study without the prior written consent of the Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03043651/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03043651/SAP_001.pdf